CLINICAL TRIAL: NCT00358657
Title: HLA-Haploidentical Related Marrow Grafts for the Treatment of Primary Immunodeficiencies and Other Nonmalignant Disorders Using Conditioning With Low-Dose Cyclophosphamide, TBI and Fludarabine and Postgrafting Cyclophosphamide
Brief Title: Fludarabine Phosphate, Cyclophosphamide, and Total-Body Irradiation Followed by Donor Bone Marrow Transplant and Cyclophosphamide, Mycophenolate Mofetil, Tacrolimus, and Sirolimus in Treating Patients With Primary Immunodeficiency Disorders or Noncancerous Inherited Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kanwaldeep K Mallhi, Assistant Professor, Clinical Research Division, Fred Hutch, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2032.00; NCI-2010-00192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2032; 2032.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01HL122173 (NIH); P30CA015704 (NIH); RG9213024 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Immunodeficiency Syndrome; Severe Aplastic Anemia; Genetic Disorder
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Anemia, Aplastic; Genetic Diseases, Inborn | interventions — Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Sirolimus; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemo, total-body irradiation, transplant) (Experimental): See Detailed Description
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Sirolimus; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic bone marrow transplantation
  Other Names: Allo BMT; Allogeneic BMT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic bone marrow transplantation
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo total-body irradiation
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase I/II trial studies the side effects of fludarabine phosphate, cyclophosphamide and total-body irradiation followed by donor bone marrow transplant and cyclophosphamide, mycophenolate mofetil, tacrolimus, and sirolimus in treating patients with primary immunodeficiency disorders or noncancerous inherited disorders. Giving low doses of chemotherapy and total-body irradiation before a bone marrow transplant helps prepare the patient's body to accept the incoming donor's bone marrow and decrease the risk that the patient's immune system will reject the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells called graft versus host disease. Giving cyclophosphamide, mycophenolate mofetil, tacrolimus, and sirolimus after the transplant may help decrease this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine safety of nonmyeloablative conditioning and hematopoietic cell transplantation (HCT) from human leukocyte antigen (HLA)-haploidentical related donors for patients with nonmalignant inherited disorders who do not have an HLA-matched related or unrelated donor.

SECONDARY OBJECTIVES:

I. Determine whether nonmyeloablative conditioning and HCT from an HLA-haploidentical related donor graft can establish mixed chimerism (> 5% cluster of differentiation [CD]3+ donor T-cell chimerism) in patients with nonmalignant inherited disorders.

II. Transplant related mortality at day 100.

III. Incidence and severity of graft-versus-host disease (GHVD).

IV. Immune reconstitution.

V. Infections during the first 200 days after HCT.

OUTLINE:

NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) over 1 hour on days -6 to -2; cyclophosphamide IV over 1 hour on days -6 and -5; and undergo total body irradiation on day -1.

TRANSPLANTATION: Patients undergo allogeneic bone marrow transplant on day 0.

POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive cyclophosphamide IV over 1 hour on days 3 and 4, and mycophenolate mofetil orally (PO) every 8 hours on days 5-30 then twice daily (BID) to day 40, and then if there is no evidence of active GVHD and donor engraftment is > 95% (or by principal investigator [PI] approval) taper until approximately day 96, or faster at discretion of PI. Patients also receive tacrolimus IV continuously over 22-24 hours starting on day 5 post-transplant and continue on tacrolimus through day 100 followed by a taper to approximately day 180 if there is no evidence of GVHD and their graft is doing well. Patients may convert to oral tacrolimus given BID or three times daily (TID) when the patient is able to take medications orally and has a therapeutic drug level. In addition, patients will receive sirolimus PO beginning on day 5 through day 180 followed by a taper to approximately day 210 if there is no evidence of GVHD and their graft is doing well.

After completion of study treatment, patients are followed up at 6, 12, 18, and 24 months, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary immunodeficiency disorder or other nonmalignant inherited disease (except Fanconi anemia) treatable by allogeneic HCT
* Patients with pre-existing medical conditions or other factors that renders them at high risk for regimen related toxicity or ineligible for conventional myeloablative HCT and who do not have HLA-matched related or unrelated donors
* Patients with a related donor who is identical for one HLA haplotype
* Acquired aplastic anemia: severe aplastic anemia (SAA) is defined as follows:

  * Bone marrow cellularity < 25%, or marrow cellularity < 50% but with < 30% residual hematopoietic cells
  * Two out of three of the following (in peripheral blood): neutrophils < 0.5 x 10^9/L; platelets < 20 x 10^9/L; reticulocytes < 20 x 10^9/L
  * SAA diagnostic criteria may be applied to assessment at initial diagnosis or follow-up assessments
* DONOR: Related donors who are identical for one HLA haplotype
* DONOR: Bone marrow will be the only allowed stem cell source

Exclusion Criteria:

* Fanconi anemia
* Suitably HLA-matched related or unrelated donors
* Patients with metabolic storage diseases who have severe central nervous system (CNS) involvement of disease, defined as intelligence quotient (IQ) score < 70
* Cardiac ejection fraction < 30% (or, if unable to obtain ejection fraction, shortening fraction < 26%) on multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (echo), symptomatic coronary artery disease, or other cardiac failure requiring therapy; patients with a history of, or current cardiac disease should be evaluated with appropriate cardiac studies and/or cardiology consult; patients with a shortening fraction of < 26% must be seen by cardiology for approval
* Poorly controlled hypertension despite anti-hypertensive medications
* Patients with clinical or laboratory evidence of liver disease will need to be evaluated for the cause of the liver disease, its clinical severity in terms of liver function and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dl, or symptomatic biliary disease
* Positive for human immunodeficiency virus (HIV)
* Females who are pregnant (beta-human chorionic gonadotropin positive [beta-HCG+]) or breast-feeding
* Fertile men or women who are unwilling to use contraceptives during HCT and up to 12 months post-treatment
* Patients with fungal pneumonia with radiological progression after receipt of amphotericin formulation or mold-active azoles for greater than 1 month will not be eligible for this protocol (either regimen A or B)
* DONOR: Donor-recipient pairs in which the HLA-mismatch is only in the host-versus-graft (HVG) direction; patients are homozygous and donor is heterozygous
* DONOR: Donors who are not expected to meet the minimum target dose of marrow cells (1 x 10^8 nucleated cells/kg recipient ideal body weight)
* DONOR: HIV-positive donors
* DONOR: A positive anti-donor cytotoxic cross match is absolute donor exclusion
* DONOR: < 6 months old and > 75 years old

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2006-05-24 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2019-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanwaldeep Mallhi, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 10.7 [0.62 to 21.45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Graft Rejection
Description: Number of patients with graft rejection (CD3 donor chimerisms <5%).
Time Frame: Day 84
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 1

2. Primary Outcome: Graft Failure
Description: Number of patients with graft failure (grade IV thrombocytopenia and neutropenia after day 21 that lasts > 2 weeks andn is refractory to growth factor support).
Time Frame: Day 84
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 0

3. Secondary Outcome: Proportion of Patients Who Achieve Greater Than 5% Donor T-cell Chimerism
Description: Number of patients who achieve greater than 5% donor T-cell (CD3+) chimerisms
Time Frame: By day 84
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 13

4. Secondary Outcome: Number of Patients With Transplant Related Mortality
Description: The number of patients with transplant related mortality
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 0

5. Secondary Outcome: Incidence of Grade I/II Acute Graft Versus Host Disease (GVHD)
Description: Number of patients diagnosed with overall GI/G2 acute GVHD by Day 100
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 7

6. Secondary Outcome: Incidence of Grade III/IV Acute Graft Versus Host Disease (GVHD)
Description: Number of patients diagnosed with overall GIII/IV acute GVHD by Day 100
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 5

7. Secondary Outcome: Incidence of Chronic GVHD
Description: Number of patients diagnosed with chronic GVHD by 1 year post transplant
Time Frame: 1 year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 11

8. Secondary Outcome: Immune Reconstitution
Description: Number of patients with normal range CD3 @ 1 year post transplant
Time Frame: 1 year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 13
Participants | 4

9. Secondary Outcome: Number of Patients With Infections
Description: Number of patients with clinically significant infections requiring treatment within 200 days after HCT
Time Frame: Through day 200 after HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
Number analyzed (Participants) | 14
Participants | 11

ADVERSE EVENTS:
Time Frame: Day 200 post initiation of conditioning therapy
Arm/Group | Treatment (Chemo, Total-body Irradiation, Transplant)
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemo, Total-body Irradiation, Transplant) (N=14)
Hypoxia requiring mechanical ventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pancreatitis with shock (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemo, Total-body Irradiation, Transplant) (N=14)
Hypotension (Vascular disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Pancreatisis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT00358657/Prot_SAP_000.pdf